CLINICAL TRIAL: NCT04275349
Title: Trial of pRehospital Intervention With trAditional Chinese Medicine for Acute strokE: A Mixed Methods Research
Brief Title: Trial of pRehospital Intervention With trAditional Chinese Medicine for Acute strokE
Acronym: TRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Beijing Emergency Medical Center (Other); Beijing Tiantan Hospital (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Centre for Evidence Based Chinese Medicine, Beijing University of Chinese Medicine (Unknown); Xuanwu Hospital, Beijing (Other); Beijing Friendship Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Fengtai Youanmen Hospital (Unknown); Beijing Jiangong Hospital (Unknown); Beijing Chaoyang Emergency Medical Center (Unknown); Beijing Chaoyang Integrative Medicine Emergency Medical Center (Unknown); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Fangshan Hospital，Beijing University of Chinese Medicine (Unknown); Civil Aviation General Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Chinese Medicine Hospital-Pinggu Hospital (Unknown); Beijing Pinggu District Hospital (Other)
Responsible Party: Principal Investigator, Ying Gao, President of the Institute for Encephalopathy, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Other Study IDs: CFH 2018-1-4191
Record Dates: First submitted 2020-02-07; First posted 2020-02-19 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Acute Ischemic Stroke; Acute Intracranial Hemorrhage
Keywords: Registry; Cohort study; Mixed methods; Prehospital; Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Exposure group(continuously): xingnaojing injection will be intravenously administered within 24 hours of symptom onset until to third day (from prehospital ambulance to hospital or at hospital)
  Interventions: Drug: Xingnaojing injection within 24 hours of symptom onset
- Exposure group(uncontinuously): xingnaojing injection will be intravenously administered within 24 hours of symptom onset for once (on prehospital ambulance )
  Interventions: Drug: Xingnaojing injection within 24 hours of symptom onset
- Completely unexposed group: xingnaojing injection will not be intravenously administered within 24 hours of symptom onset until to third day (from prehospital ambulance to hospital)
- Incompletely unexposed group: xingnaojing injection will not be intravenously administered on ambulance but administered more than 24 hours of symptom onset at hospital

INTERVENTIONS:
Drug: Xingnaojing injection within 24 hours of symptom onset — intravenously administered Xingnaojing injection within 24 hours of symptom onset on ambulance or at hospital
  Groups: Exposure group(continuously); Exposure group(uncontinuously)

SUMMARY:
The main purpose of this trial is to observe whether Xingnaojing, intravenously administered within 24 hours of symptom onset on pre-hospital emergency ambulance, improves the Early neurological deterioration of acute stroke at 3 days.

DETAILED DESCRIPTION:
The TRACE is a multicenter, registry observational study. Xingnaojing injection is the only essential traditional chinese medicine on emergency ambulance used for acute stroke.The primary hypothesis of this trial is that Xingnaojing used for acute stroke within 24 hours of symptom onset on ambulance will improve the Early neurological deterioration of acute stroke at 3 days. All suspected acute stroke participants will be registered once they are taken on the ambulance. The primary outcome will be determined at 3 days.Besides, there will be a quantitative interview with emergency doctors about their knowledge and attitude on Xingnaojing for acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of suspected acute stroke；
* Symptom onset within 24 hours；
* Age ≥ 18 .

Exclusion Criteria:

* Other conditions that lead to motor dysfunction (e.g., severe osteoarthrosis, rheumatoid arthritis);
* Other conditions that render outcomes or follow-up unlikely to be assessed; Known to be pregnant or breastfeeding;
* Non-acute stroke (result from Computed Tomography(CT) or Magnetic Resonance Imaging(MRI)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: suspected acute stroke patient (call for emergency ambulance)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Early neurological deterioration（change between baseline and 3 days) | 3 days
  The early neurologic deterioration is defined as an increase of 1 points or more in the National Institute of Health Stroke Scale (NIHSS) score between baseline and 3 days. The NIHSS score ranges from 0 (best score) to 42 (worst score).

SECONDARY OUTCOMES:
Rate of stroke related deaths and deaths from any cause | 14 days during hospitalization
  Rate of stroke related deaths and deaths from any cause during hospitalization
Neurological impairment | Baseline and day of discharge or 10 days
  Evaluated by National Institute of Health Stroke Scale (NIHSS)
Risk grade of cerebral hemorrhage | Baseline and day of discharge or 10 days
  Intracranial hemorrhage evaluated by Intracerebral Haemorrhage(ICH) scale.
Activities of daily living | 30 days,60 days and 90 days
  Activities of daily living will be measured by Barthel Index (BI)score at 30 days and 90 days.The Barthel Index score ranges from 0 (worst score) to 100 (best score).
The proportion of patients independent | 30 days,60 days and 90 days
  The proportion of patients independent will be evaluated by modified Rankin Scale(mRS).The mRS score ranges from 0 (best score) to 6 (worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Y, Tian Z, Wang S, Liu H, Liu Y, Peng W, Lai X, Qi D, Kong L, Gao Y. Trial of a prehospital intervention with traditional Chinese medicine for acute stroke (TRACE): Protocol for a mixed-methods research study. Front Pharmacol. 2022 Aug 29;13:879282. doi: 10.3389/fphar.2022.879282. eCollection 2022. PMID 36105230